# Effects of Pioglitazone on Stress Reactivity and Alcohol Craving NCT03860753

Version Date: 05/08/2019

## **ABSTRACT**

Alcohol use disorder (AUD) is associated with significant negative health, social, and economic costs. Alcohol activates the hypothalamic-pituitary-adrenocortical (HPA)-axis, and stress can increase the reward value of drinking. Continued excessive drinking results in behavioral changes marked by increased compulsive drinking, stress reactivity, and neuro-inflammation<sup>8</sup>. FDA-approved pharmacotherapies for AUD (e.g., naltrexone, acamprosate, disulfiram) are effective in less than a third of treated individuals<sup>9</sup>. *Importantly, none of the currently approved medications for AUD directly address stress reactivity, underscoring the need to develop novel pharmacotherapies targeting stress-related processes associated with AUD.* 

A promising pharmacological target for addressing AUD and stress reactivity is the family of peroxisome proliferator-activated receptors (PPARs), proteins that act as ligand-activated transcription factors that exhibit both anti-inflammatory and neuro-protective responses in the brain¹o. A growing number of pre-clinical models have shown promising effects of PPAR agonists on drug-related outcomes¹¹. For example, the PPARγ agonist pioglitazone 1) significantly reduced free-access alcohol consumption; and 2) attenuated alcohol consumption and withdrawal symptoms following stress exposure in rats bred to highly prefer alcohol¹²,¹³. An important innovation of the current study will be to translate these results for the first time to humans with AUD.

The primary purpose of the current proposal is to obtain preliminary data to increase the likelihood of funding for a future NIH grant, while balancing the feasibility of completing the current proposal. To that end, we will utilize a within-subject, repeated measures design to assess the feasibility of administering pioglitazone for four weeks to non-treatment and treatment-seeking individuals with AUD and elevated levels of stress/anxiety (N=20). Participants will undergo pre- and post-treatment human laboratory assessment of stress-reactivity and stress-induced alcohol craving. During treatment, changes in alcohol use, stress/anxiety, and alcohol craving will be assessed in the natural environment. The study design features 1) rigorous monitoring of medication compliance (Medication Event Monitoring System (MEMs)) and alcohol use (urinary ethyl glucuronide (ETG)); 2) biological assessment of stress reactivity (salivary cortisol, blood pressure, and heart rate); and 3) a multi-dimensional assessment of stress-induced alcohol craving incorporating both traditional measures of alcohol craving in addition to relatively novel behavioral economic measures (delay discounting, alcohol demand). Taking these measures together, we hope to present a robust and comprehensive characterization of pioglitazone on alcohol use, stress reactivity, and stress-induced alcohol craving.

# **SPECIFIC AIMS**

**Specific Aim 1:** To assess pre- to post-treatment reductions in stress reactivity (self-report, salivary cortisol, heart rate, blood pressure) and stress-induced alcohol craving (self-report, alcohol demand) in the human laboratory setting.

*Hypothesis* 1: We will observe pre- to post- treatment reductions in stress reactivity and stress-induced alcohol craving.

**Specific Aim 2:** To assess changes in alcohol drinking (drinks per day, heavy drinking days), stress/anxiety (PSS, HAMA, PCL-5), and alcohol craving (PACS, delay discounting, alcohol demand) during treatment in the natural environmental setting.

**Hypothesis 2:** We will observe decreased alcohol drinking, stress/anxiety, and alcohol craving over the course of treatment.

There is increasing attention and evidence supporting the potential role of the PPARy system as a novel target in the treatment of AUD. From a translational perspective, this study is timely and likely to advance our understanding of stress as a mechanism of action of pioglitazone effects.

IRB NUMBER: HSC-MS-18-0922

UTHealth IRB APPROVAL DATE: 05/08/2019

#### BACKGROUND AND RATIONALE

<u>Public Health Impact of AUD.</u> AUD is 1) the 4<sup>th</sup> leading cause of death in the US (~88,000 deaths/year), decreasing lifespan by approximately 30 years; 2) a tremendous economic burden on society (~\$249 billion/year); and 3) associated with a host of short- and long-term negative consequences including violence, legal problems, morbidity, and family problems<sup>14–16</sup>.

AUD and the Central Role of Stress. Persistent excessive drinking is a chronic stressor that 1) shifts brain systems beyond normal homeostatic limits into a state of allostasis; 2) which in turn alters physiological and brain motivational systems central for regulating alcohol use; and 3) has negative impact on autoimmune and inflammatory responses that can in turn influence alcohol use<sup>17–21</sup>. Whereas initial drinking is influenced by the positive reinforcing effects of alcohol and impulsivity, continued drinking adopts compulsive characteristics maintained increasingly by negative reinforcement (e.g., alcohol withdrawal symptoms, stress-related anxiety, alcohol craving) as well as decreased stress-resiliency and cognitive deficits from neuro-inflammatory damage<sup>17,22,23</sup>. Despite the profound negative impact of stress on AUD, *none of currently approved medications for AUD directly target stress or stress-related consequences associated with AUD*.

Novelty and Promise of the PPAR System. PPARs are proteins that act as ligand-activated transcription factors, which is central to their anti-inflammatory actions<sup>24</sup>. Pre-clinical studies highlight the potential of PPAR agonists on various aspects of drug use (e.g., discrimination, self-administration, reinstatement, sensitization) for several drugs of abuse including alcohol<sup>11</sup>. In human studies, expression of PPAR has been shown to be altered among individuals with AUD in genome-wide association studies (GWAS) <sup>25</sup> studies. In a recent study by our group, post hoc analyses revealed significantly decreased alcohol use among individuals with concurrent cocaine use disorder (CUD) and AUD receiving the PPARγ agonist pioglitazone, compared to placebo, in a study assessing cocaine craving and white matter integrity.<sup>27</sup>.

Currently, only the PPAR gamma (PPARy) isoform can be targeted in humans. PPARy is highly expressed in a number of brain regions associated with drug reward<sup>28</sup> and stress response<sup>12,13</sup>. Activation of PPARy mediates neuroprotective responses against inflammatory damage, which can attenuate drug affects<sup>29–32</sup>. The PPARy agonist Pioglitazone (Actos) is FDA-approved for the treatment of diabetes and metabolic disorders. In preclinical studies, pioglitazone protects against 1) alcohol-induced neuronal and cognitive damage in a model of binge-drinking<sup>33</sup>; and 2) neuro-inflammation and neurodevelopmental toxicity in a model of fetal alcohol spectrum disorder<sup>34</sup>. Directly relevant to the current study, *pioglitazone 1*) *significantly reduced alcohol drinking in rats; and 2*) attenuated stress-induced alcohol drinking and alcohol withdrawal symptoms in rats bred to highly prefer alcohol<sup>12,13</sup>.

Multi-Dimensional Assessment of Alcohol-Induced Craving. Self-report measures of drug craving are ubiquitous and often serves as a proxy of motivation to consume drug but have limitations that have likely resulted in equivocal results in human laboratory studies<sup>35</sup>. Behavioral economic measures (i.e., delay discounting, alcohol demand) may help mitigate these issues and are both closely associated with drug use and directly tied to a broader framework of drug addiction. Delay discounting is a relatively stable, trait-like measure that assesses the decrease in value of a reward as a function to delay of its receipt, and also serves as a measure of impulsivity. Delay discounting has an extensive literature revealing associations with virtually every aspect of drug use including initiation, severity, and relapse risk<sup>36–38</sup>. Alcohol demand assesses how much alcohol an individual is willing to consume as a function of increasing price, serving as 1) a robust characterization of the reward value of alcohol and therefore craving; and 2) a proxy of compulsive drug use (i.e., consuming alcohol despite increasing aversive consequences). Drug demand can be easily and quickly assessed through purchasing tasks, which have very strong reliability, predictive validity, and are sensitive to state-dependent changes in demand under conditions of withdrawal, cue exposure, environmental stressors,

IRB NUMBER: HSC-MS-18-0922 UTHealth IRB APPROVAL DATE: 05/08/2019 and predict alcohol treatment response<sup>39–42</sup>. Delay discounting and alcohol demand are poorly correlated with each other, supporting a multi-dimensional model in which these measures represent distinct aspects of motivation to use alcohol<sup>42–48</sup>. In the current proposal, we will assess changes in both delay discounting and alcohol demand over Study Weeks o to 4 and alcohol demand will be used to assess state-dependent changes during the human laboratory stress-reactivity assessment.

## **METHODS**

**Research team.** The research team will consist of Dr. Yoon (PI) and a number of collaborators from UTHealth and Brown University. Dr. Yoon (PI) is an experienced addiction researcher and an expert in assessing behavioral economic measures in addiction research, which is pertinent to the current project. Drs. Weaver (CNRA Medical Director) and Lin (Addictions Psychiatrist) will provide medical guidance and ensure participant safety over the course of the study. Dr. Lane is Professor and Vice Chair for Research and directs the Behavioral Laboratory at the CNRA with expertise in medication development trials as well as alcohol studies. Dr. Suchting is a biostatistician and data scientist with expertise in experimental design and statistical modeling, including the type of generalized linear modeling that will be utilized by the present research. From Brown University, Dr. Haas-Koffler (Co-I) is serving as a consultant on this project and is an expert in stress and alcohol research<sup>1-7</sup>. Additionally, our group has a history of collaborating with the Laboratory of Biomarkers located in the BBSB for analyzing biological samples, such as salivary cortisol in the current protocol. We will work with Dr. Fries to ensure that samples are collected and analyzed appropriately.

<u>Overall study design.</u> We will utilize a within-subject, repeated measures design. Participants will receive pioglitazone or placebo for four weeks. A summary of the study timeline, procedures, and assessments is shown in the following Table.

Table 1. Outline of Study Timeline, Procedures, and Assessments

| Study Week | 0 | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|
| Procedures and Assessments | | | | | |
| Consent and Baseline Screening | | | | | |
| SCID, ASI, KMSK, TLFB, CIWAA, AUDIT | X | | | | |
| Receive Study Medication (Pioglitazone or Placebo) | X | X | X | X | |
| Assess Medication Compliance and Adverse Events | | X | X | X | X |
| Human Laboratory Procedures (Specific Aim 1) | | | | | |
| Stress-Reactivity Assessment (Salivary Cortisol, HR, BP, Craving) | X | | | | X |
| Alcohol Demand, Alcohol Ladder | X | | | | X |
| Natural Environment Procedures (Specific Aim 2) | | | | | |
| Alcohol Use and Craving (Self-Report, BrAC, ETG, PACS) | X | X | X | X | X |
| Stress and Anxiety (HAM-A, PSS, BDI-II, PCL-5) | X | X | X | X | X |
| Delay Discounting, Alcohol Demand | X | X | X | X | X |

SCID - Structured Clinical Interview for DSM-5, **ASI** - Addiction Severity Index<sup>49</sup>; KMSK - Kreek-McHugh-Schluger-Kellogg scale<sup>50</sup>; **TLFB** - Timeline Followback<sup>51</sup>; CIWAA - Clinical Institute Withdrawal Assessment for Alcohol<sup>52</sup>; **AUDIT** - Alcohol Use Identification Test<sup>53</sup>; **BrAC** - Breath Alcohol Concentration; **ETG** - Ethyl Glucuronide; **PACS** - Pennsylvania Alcohol Craving Scale<sup>54</sup>; **HR** - Heart Rate; **BP** - Blood Pressure; **HAM-A** - Hamilton Anxiety Rating Scale<sup>55</sup>; **PSS** - Perceived Stress Scale<sup>56</sup>; **PCL-5** - PTSD Checklist for DSM-5; **BDI-II** - Beck Depression Inventory - II.

**Participants, Recruitment, and Setting.** Participants **(N=20)** will consist of non-treatment and treatment-seeking individuals diagnosed with AUD (DSM-5) between 21 to 40 years old and fluent in English; past month excessive alcohol use (>7 drinks/week for woman, >14 drinks/week for men, >3 drinks/occasion for women>4 drinks/occasion for men)<sup>14</sup>; baseline HAM-A or PSS Score indicative of mild to moderate anxiety (score 8 to 23) or moderate stress (score 14 to 26), respectively; and increase in alcohol straying following the 0922

baseline stress reactivity assessment. Individuals will be excluded for exhibiting severe scores on the HAM-A, PSS, BDI-II, or PTSD checklist (PCL-5) at the discretion of the admitting physician (Dr. Weaver); physical dependence on alcohol; greater than mild substance use disorder on drugs other than alcohol, nicotine, and marijuana; contraindications for taking pioglitazone; medical conditions contraindicating pioglitazone pharmacotherapy or taking contraindicated medications; be pregnant, nursing, or planning on becoming pregnant during the course of the study; have any other illness, condition, or use of medications, which in the opinion of the PI and/or admitting physician would preclude safe and/or successful completion of the study. Recruitment strategies will include local advertising in print media, public service announcements on radio, and referrals to CNRA in the Houston metropolitan area.

**Baseline Screening.** Participants will receive a comprehensive medical and psychiatric evaluation including: a medical-history questionnaire, physical examination, laboratory chemistries (e.g., blood chemistry screen, complete blood count, urinalysis and urine pregnancy test), and ECG. Clinicians will conduct the **SCID**, the **ASI** ASI<sup>49</sup>, the **KMSK**<sup>50</sup> assessment of lifetime substance use interview, and **TLFB**<sup>51</sup>. Alcohol dependence will be assessed using the SCID and the **CIWAA**<sup>52</sup>.

Alcohol-Related Measures. Assessment of alcohol use will include self-report (TLFB), BrAC (Alco-Sensor FST, Intoximeters, Inc., Saint Louis, MO). Severity of alcohol use will be assessed using the AUDIT<sup>53</sup>. Motivation to quit will be assessed using the Alcohol Ladder questionnaire. Alcohol craving will be assessed using a 5-item questionnaire<sup>57</sup>. ETG will be assessed using dipcards with a 300 ng/ml cutoff. ETG dipcards show good agreement with traditional immunoassays<sup>58-60</sup>.

Behavioral Economic Measures. Alcohol demand will be assessed via the Brief Assessment of Alcohol Demand (BAAD)<sup>42</sup>, a 3-item questionnaire measuring the three most common indices of alcohol demand. Delay discounting will be assessed for both money and alcohol using a computerized task at weekly clinic visits developed by Dr. Yoon (PI)<sup>61,62,71,63–70</sup>.

**Stress and Anxiety Measures.** Stress and anxiety levels will be assessed using the **HAM-A**<sup>55</sup>, **PSS**<sup>56</sup>, **BDI-II**, and the **PCL-5**. Established norms will be used for the HAM-A and PSS to assess mild to moderate stress and anxiety and screen out for cases of severe stress and anxiety.

<u>Stress Reactivity Measures.</u> HR and BP will be assessed using standard laboratory equipment. Saliva samples will be collected in swabs using the Cortisol-Salivette® system (Sarstedt) and measured using the Cortisol ELISA Kit (Enzo Life Sciences), per manufacture instructions.

Study Medication. Pioglitazone (Actos®, Takeda Pharmaceuticals U.S.A., Inc.) is FDA-approved for the treatment of diabetes mellitus type 2; has anti-inflammatory, neuroprotective, antioxidative, and anti-excitotoxic properties<sup>72</sup>; and extensive research has shown it to be safe in human patient populations<sup>73,74</sup>. The medication schedule is based on previous work from our group showing that a daily dose of 45mg was associated with acceptable levels of tolerability, safety, and compliance in a study assessing the effects of pioglitazone on individuals with CUD and AUD<sup>27</sup>. Our pilot trial used a conservative 2-week dose titration schedule (i.e., Week 1: 15 mg/d; Week 2: 30 mg/d), with no adverse effects reported or observed. For the current trial we will follow recommended adult initial dosing at 30 mg/d to reach maintenance dose of 45 mg/d by week 2, which is within standard titration parameters as per the investigator's brochure. Thorough screening of all subjects including history and physical examination, serum chemistry and hematology, EKG, urinalysis and Urine Drug Screen as well as structured psychiatric interviews will be completed on all subjects. Exclusion criteria include subjects at greatest risk of side effects of pioglitazone, including those with congestive heart failure, significant liver disease, edema, and diabetes, as well as risks of alcohol use (pregnant IRB NUMBER: HSC-MS-18-0922

IRB NUMBER: HSC-MS-18-0922
UTHealth
IRB APPROVAL DATE: 05/08/2019

women). Monitoring of weight to capture potential fluid retention will occur at each visit along with an adverse event assessment to include assessment for edema. Blood will be drawn at the end of the study for liver function testing. Female subjects must agree to use an effective barrier method of birth control and urine pregnancy tests will be performed at each visit to minimize risk of pregnancy.

Medication Compliance. One week supplies of the study medication will be dispensed with a Medication Event Monitoring System (MEMS) cap to record the number of bottle openings and date/time of each opening. Riboflavin will be added to medication capsules and urine ultraviolet fluorescent tests will be conducted at weekly clinic visits to assess compliance. Participants will receive \$10 at each clinic visit in which results from self-report, MEMS, and riboflavin are all consistent with medication compliance.

Human Laboratory Procedures (Specific Aim 1). On Study Weeks 0 and 4, participants will engage in the cold-pressor task (CPT). The CPT is widely used as a stress-inducer in human laboratory studies and elicits moderate activation of the sympathetic nervous system and limited activation of the HPA-axis, which are two major stress systems in the body<sup>75–78</sup>. HPA-axis activation during the CPT can be increased by

incorporating a social evaluative component. Specifically, a study member of the opposite sex of the study participant will dress in a white labcoat and be physically present during the CPT. Additionally, participants will be videotaped and informed that their facial expressions will be assessed during the CPT. The addition of the social component during the CPT has been demonstrated to selectively activate the HPA-axis and significantly increase salivary cortisol levels<sup>77</sup>. During the CPT, participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Stress levels will be assessed using subjective and physiological measures HR, BP, and salivary cortisol consistent with previous studies from our group<sup>79,80</sup>. Alcohol craving will be assessed using a 4-item questionnaire<sup>57</sup>.

Table 2. Time Course for Assessing Stress-Induced Relapse Risk

| Time | Study |
|------|--------------------------|
| (pm) | Procedures |
| 3:00 | Assess Craving, BAAD, |
| | Stress, Cortisol, HR, BP |
| 3:15 | Cold Pressor Task |
| 3:20 | Assess Craving, BAAD, |
| | Stress, HR, BP |
| 3:45 | Assess Craving, BAAD, |
| | Stress, Cortisol, HR, BP |

Natural Environment Procedures (Specific Aim 2). At Study Week o, all participants will receive a pamphlet copy of the "Rethinking Drinking: Alcohol and Your Health" providing research-based information related to alcohol use (Rethinking Drinking.niaaa.nih.gov). Research staff will go over the pamphlet's information with the participant at the initial visit and subsequent visits as necessary. At each study visit, participants will receive study medication for the week and assessed for adverse events and medication compliance. At each visit, participants will also be assessed for recent alcohol use (self-report, ETG, BrAC), alcohol craving (PACS), and stress/anxiety (HAM-A, PSS). At the end of the study, participants will be referred to local alcohol treatment services as needed.

<u>Participant Payment & Compensation.</u> Participants will receive be able to receive \$300 for completing the study (\$50 for completing baseline screening; \$25 for each visit (\$100); \$25 for stress reactivity assessments (\$50); and \$100 completion bonus). Additionally, participants will potentially receive \$10/week (up to \$40) for demonstrating medication compliance. Participants will also receive parking/bus fare compensation at each visit worth \$5.

# **DATA ANALYSIS PLAN**

**General Data Analytic Strategy.** Analyses will proceed in parallel using frequentist and Bayesian statistical inference. Frequentist analyses will examine relationships between predictors and outcomes using traditional measures of effect size and statistical significance (i.e., regression coefficients, standard errors, IRB NUMBER: HSC-MS-18-0922

UTHealth IRB APPROVAL DATE: 05/08/2019

confidence intervals, and p-values), while Bayesian analyses will measure uncertainty in model parameter estimates via posterior distributions and directly evaluate the probability of the alternative hypothesis.

**Specific Aim 1**: assess pre- to post-treatment reductions in stress reactivity (self-report, salivary cortisol, heart rate, blood pressure) and stress-induced alcohol craving (self-report, alcohol demand) in the human laboratory setting.

Hypothesis 1: We will observe pre- to post- treatment reductions in stress reactivity and stress-induced alcohol craving. Generalized linear mixed modeling will be used to evaluate each outcome as a function of time (pre-test and post-test) in unique models.

**Specific Aim 2:** Demonstrate reduced alcohol drinking (drinks per day, heavy drinking days), stress/anxiety (PSS, HAMA, PCL-5), and alcohol craving (PACS, delay discounting, alcohol demand) during treatment in the natural environmental setting.

Hypothesis 2: We will observe decreased alcohol drinking, stress/anxiety, and alcohol craving over the course of treatment. Generalized linear mixed modeling will be used to evaluate each outcome as a function of time in unique models. Alcohol consumption will be modeled via drinks per drinking day, such that the number of positive drinking episodes a participant experienced in a week will be included as a count outcome (i.e., Poisson-distributed) and the number of drinking days in a week will be controlled for as an off-set covariate.

**Power/Sample Size Considerations.** The frequentist framework using null hypothesis statistical testing can provide some understanding of changes over time for each outcome. However, in evaluating a small within-subjects pilot trial of N = 20 participants, Bayesian statistical inference provides a superior framework for deriving evidence regarding the magnitude and direction of change over time for each model. The posterior probability of each effect would then be useful to inform effect sizes for power calculations and/or prior distributions in future research. As due diligence, however, a conventional frequentist power analysis follows. For the current proposal, power estimates are calculated using G\*Power 3.1.9.2 and focus on reduction in alcohol consumption. Assuming alpha = 0.05 (one-tailed), an average baseline rate of 10.5 drinks/week across all participants (averaged between 14 and 7 drinks/week for male and female participants, respectively), a sample size of N = 20 participants provides 80% power to detect a 20% decrease in alcohol consumption over five weeks.



IRB NUMBER: HSC-MS-18-0922 UTHealth IRB APPROVAL DATE: 05/08/2019

## **REFERENCES**

- 1. Haass-Koffler CL, Leggio L, Kenna GA. Pharmacological approaches to reducing craving in patients with alcohol use disorders. *CNS Drugs*. 2014;28(4):343-360. doi:10.1007/s40263-014-0149-3
- 2. Kenna GA, Haass-Koffler CL, Zywiak WH, et al. Role of the alpha1 blocker doxazosin in alcoholism: a proof-of-concept randomized controlled trial. *Addict Biol.* 2016;21(4):904-914. doi:10.1111/adb.12275
- 3. Haass-Koffler CL, Henry AT, Melkus G, et al. Defining the role of corticotropin releasing factor binding protein in alcohol consumption. *Transl Psychiatry*. 2016;6(11):e953. doi:10.1038/tp.2016.208
- 4. Haass-Koffler CL, Bartlett SE. Stress and addiction: contribution of the corticotropin releasing factor (CRF) system in neuroplasticity. *Front Mol Neurosci.* 2012;5:91. doi:10.3389/fnmol.2012.00091
- 5. K. G, C.L. H-K, S.E. E, et al. Elasticity of alcohol demand as a moderator of alcohol drinking in alcohol-dependent individuals treated with doxazosin. *Alcohol Clin Exp Res.* 2017. doi:http://dx.doi.org/10.1111/acer.13391
- 6. M. F, C. H-K, W. Z, R.M. S, G.A. K. Noradrenergic system as a pharmacological target for alcoholism: A randomized, double-blind, placebo-controlled, proof-of-concept, clinical trial with doxazosin. *Biol Psychiatry*. 2015.
- 7. C.L. H-K, L. L. The alpha1 blockade by doxazosin in regulation of alcohol drinking in alcohol dependent patients. *Alcohol Clin Exp Res.* 2017. doi:http://dx.doi.org/10.1111/acer.13392
- 8. Kwako LE, Koob GF. Neuroclinical Framework for the Role of Stress in Addiction. *Chronic Stress* (*Thousand Oaks*). 2017;1. doi:10.1177/2470547017698140
- 9. Miller G. Psychopharmacology. Tackling alcoholism with drugs. *Science* (80- ). 2008;320(5873):168-170. doi:10.1126/science.320.5873.168
- 10. Munhoz CD, Garcia-Bueno B, Madrigal JL, Lepsch LB, Scavone C, Leza JC. Stress-induced neuroinflammation: mechanisms and new pharmacological targets. *Braz J Med Biol Res*. 2008;41(12):1037-1046. https://www.ncbi.nlm.nih.gov/pubmed/19148364.
- 11. Le Foll B, Di Ciano P, Panlilio L V, Goldberg SR, Ciccocioppo R. Peroxisome proliferator-activated receptor (PPAR) agonists as promising new medications for drug addiction: preclinical evidence. *Curr Drug Targets*. 2013;14(7):768-776. https://www.ncbi.nlm.nih.gov/pubmed/23614675.
- 12. Stopponi S, de Guglielmo G, Somaini L, et al. Activation of PPARgamma by pioglitazone potentiates the effects of naltrexone on alcohol drinking and relapse in msP rats. *Alcohol Clin Exp Res.* 2013;37(8):1351-1360. doi:10.1111/acer.12091
- 13. Stopponi S, Somaini L, Cippitelli A, et al. Activation of nuclear PPARgamma receptors by the antidiabetic agent pioglitazone suppresses alcohol drinking and relapse to alcohol seeking. *Biol Psychiatry*. 2011;69(7):642-649. doi:10.1016/j.biopsych.2010.12.010
- 14. Centers for Disease Control and Prevention. Fact Sheets Alcohol Use and Your Health. https://www.cdc.gov/alcohol/fact-sheets/alcohol-use.htm. Published 2016.
- 15. Sacks JJ, Gonzales KR, Bouchery EE, Tomedi LE, Brewer RD. 2010 National and State Costs of Excessive Alcohol Consumption. *Am J Prev Med.* 2015;49(5):e73-9. doi:10.1016/j.amepre.2015.05.031
- 16. Stahre M, Roeber J, Kanny D, Brewer RD, Zhang X. Contribution of excessive alcohol consumption to deaths and years of potential life lost in the United States. *Prev Chronic Dis.* 2014;11:E109. doi:10.5888/pcd11.130293
- 17. Koob G, Kreek MJ. Stress, dysregulation of drug reward pathways, and the transition to drug dependence. *Am J Psychiatry*. 2007;164(8):1149-1159. doi:10.1176/appi.ajp.2007.05030503
- 18. Koob GF. A role for brain stress systems in addiction. *Neuron*. 2008;59(1):11-34. doi:10.1016/j.neuron.2008.06.012
- 19. Koob GF. Brain stress systems in the amygdala and addiction. *Brain Res.* 2009;1293:61-75. doi:10.1016/j.brainres.2009.03.038
- 20. Sinha R. How does stress increase risk of drug abuse and relapse? *Psychopharmacol*. 2001;158(4):343-359. doi:10.1007/s002130100917
- 21. Sinha R. How does stress lead to risk of alcohol relapse? *Alcohol Res.* 2012;34(4):432-440. http://www.ncbi.nlm.nih.gov/pubmed/23584109.
- 22. McEwen BS, Gianaros PJ. Central role of the brain in stress and adaptation: links to socioeconomic status, health, and disease. *Ann N Y Acad Sci.* 2010;1186:190-222. doi:10.1111/j.1749-6632.2009.05331.x
- 23. Valdez GR, Koob GF. Allostasis and dysregulation of corticotropin-releasing factor and neuropeptide Y systems: implications for the development of alcoholism. *Pharmacol Biochem Behan* 3004;79(4):6781-0922

- 689. doi:10.1016/j.pbb.2004.09.020
- 24. Daynes RA, Jones DC. Emerging roles of PPARs in inflammation and immunity. *Nat Rev Immunol*. 2002;2(10):748-759. doi:10.1038/nri912
- 25. Ponomarev I, Wang S, Zhang L, Harris RA, Mayfield RD. Gene coexpression networks in human brain identify epigenetic modifications in alcohol dependence. *J Neurosci.* 2012;32(5):1884-1897. doi:10.1523/JNEUROSCI.3136-11.2012
- 26. Blednov YA, Benavidez JM, Black M, et al. Peroxisome proliferator-activated receptors alpha and gamma are linked with alcohol consumption in mice and withdrawal and dependence in humans. *Alcohol Clin Exp Res.* 2015;39(1):136-145. doi:10.1111/acer.12610
- 27. Schmitz JM, Green CE, Hasan KM, et al. PPar-gamma agonist pioglitazone modifies craving intensity and brain white matter integrity in patients with primary cocaine use disorder: A pilot trial of target assessment. *Addiction*. 2017;112(10):1861-1868. doi:10.1111/add.13868
- 28. Ubaldi M, Cannella N, Ciccocioppo R. Emerging targets for addiction neuropharmacology: From mechanisms to therapeutics. *Prog Brain Res.* 2016;224:251-284. doi:10.1016/bs.pbr.2015.07.018
- 29. Berger J, Moller DE. The mechanisms of action of PPARs. *Annu Rev Med.* 2002;53:409-435. doi:10.1146/annurev.med.53.082901.104018
- 30. Kapadia R, Yi JH, Vemuganti R. Mechanisms of anti-inflammatory and neuroprotective actions of PPAR-gamma agonists. *Front Biosci*. 2008;13:1813-1826. http://www.ncbi.nlm.nih.gov/pubmed/17981670.
- 31. Landreth GE, Heneka MT. Anti-inflammatory actions of peroxisome proliferator-activated receptor gamma agonists in Alzheimer's disease. *Neurobiol Aging*. 2001;22(6):937-944. http://www.ncbi.nlm.nih.gov/pubmed/11755002.
- 32. Tontonoz P, Spiegelman BM. Fat and beyond: the diverse biology of PPARgamma. *Annu Rev Biochem*. 2008;77:289-312. doi:10.1146/annurev.biochem.77.061307.091829
- 33. Cippitelli A, Domi E, Ubaldi M, et al. Protection against alcohol-induced neuronal and cognitive damage by the PPARgamma receptor agonist pioglitazone. *Brain Behav Immun*. 2017;64:320-329. doi:10.1016/j.bbi.2017.02.001
- 34. Komada M, Hara N, Kawachi S, et al. Mechanisms underlying neuro-inflammation and neurodevelopmental toxicity in the mouse neocortex following prenatal exposure to ethanol. *Sci Rep.* 2017. doi:10.1038/s41598-017-04289-1
- 35. Tiffany ST, Conklin CA. A cognitive processing model of alcohol craving and compulsive alcohol use. *Addiction*. 2000;95 Suppl 2:S145-53. http://www.ncbi.nlm.nih.gov/pubmed/11002909.
- 36. Madden GJ, Bickel WK. Impulsivity: The Behavioral and Neurological Science of Discounting. 2010.
- 37. Amlung M, Vedelago L, Acker J, Balodis I, MacKillop J. Steep delay discounting and addictive behavior: a meta-analysis of continuous associations. *Addiction*. 2017;112(1):51-62. doi:10.1111/add.13535
- 38. MacKillop J, Tidey JW. Cigarette demand and delayed reward discounting in nicotine-dependent individuals with schizophrenia and controls: An initial study. *Psychopharmacology (Berl)*. 2011;216(1):91-99. doi:10.1007/s00213-011-2185-8
- 39. Amlung M, MacKillop J. Understanding the effects of stress and alcohol cues on motivation for alcohol via behavioral economics. *Alcohol Clin Exp Res.* 2014;38(6):1780-1789. doi:10.1111/acer.12423
- 40. Amlung MT, Acker J, Stojek MK, Murphy JG, MacKillop J. Is talk "cheap"? An initial investigation of the equivalence of alcohol purchase task performance for hypothetical and actual rewards. *Alcohol Clin Exp Res.* 2012;36(4):716-724. doi:10.1111/j.1530-0277.2011.01656.x
- 41. MacKillop J, O'Hagen S, Lisman SA, et al. Behavioral economic analysis of cue-elicited craving for alcohol. *Addiction*. 2010;105(9):1599-1607. doi:10.1111/j.1360-0443.2010.03004.x
- 42. Owens MM, Murphy CM, MacKillop J. Initial Development of a Brief Behavioral Economic Assessment of Alcohol Demand. *Psychol Conscious (Wash D C)*. 2015;2(2):144-152. doi:10.1037/cns0000056
- 43. Acker J, MacKillop J. Behavioral economic analysis of cue-elicited craving for tobacco: a virtual reality study. *Nicotine Tob Res.* 2013;15(8):1409-1416. doi:10.1093/ntr/nts341
- 44. MacKillop J, Brown CL, Stojek MK, Murphy CM, Sweet L, Niaura RS. Behavioral economic analysis of withdrawal- and cue-elicited craving for tobacco: an initial investigation. *Nicotine Tob Res*. 2012;14(12):1426-1434. doi:10.1093/ntr/nts006
- 45. MacKillop J, Few LR, Murphy JG, et al. High-resolution behavioral economic analysis of cigarette demand to inform tax policy. *Addiction*. 2012;107(12):2191-2200. doi:10.1111/j.1360-0443.2012.03991.x
- 46. Mackillop J, Menges DP, McGeary JE, Lisman SA. Effects of craving and DRD4 VNTR genotype on the

  IRB NUMBER: HSC-MS-18-0922

IRB NUMBER: HSC-MS-18-0922
UTHealth
The University of Texas
IRB APPROVAL DATE: 05/08/2019

- relative value of alcohol: an initial human laboratory study. *Behav Brain Funct*. 2007;3:11. doi:10.1186/1744-9081-3-11
- 47. MacKillop J, Miranda Jr. R, Monti PM, et al. Alcohol demand, delayed reward discounting, and craving in relation to drinking and alcohol use disorders. *J Abnorm Psychol*. 2010;119(1):106-114. doi:10.1037/a0017513
- 48. McKee SA, O'Malley SS, Shi J, Mase T, Krishnan-Sarin S. Effect of transdermal nicotine replacement on alcohol responses and alcohol self-administration. *Psychopharmacol*. 2008;196(2):189-200. doi:10.1007/s00213-007-0952-3
- 49. McLellan AT, Kushner H, Metzger D, et al. The fifth edition of the addiction severity index. *J Subst Abuse Treat*. 1992. doi:10.1016/0740-5472(92)90062-S
- 50. Kellogg SH, McHugh PF, Bell K, et al. The Kreek-McHugh-Schluger-Kellogg scale: A new, rapid method for quantifying substance abuse and its possible applications. *Drug Alcohol Depend*. 2003. doi:10.1016/S0376-8716(02)00308-3
- 51. Sobbell LC, Sobell MB. *Alcohol Timeline Followback Users' Manual*. Toronto, Canada: Addiction Research Foundation; 1995.
- 52. Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). *Br J Addict*. 1989;84(11):1353-1357. https://www.ncbi.nlm.nih.gov/pubmed/2597811.
- 53. Babor TF, Higgins-Biddle JC, Saunders JB, Monteiro MG. The Alcohol Use Disorders Identification Test Guidelines for Use in Primary Care. In: *World Health Organization*.; 2001. doi:10.1177/0269881110393051
- 54. Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. *Alcohol Clin Exp Res.* 1999;23(8):1289-1295. https://www.ncbi.nlm.nih.gov/pubmed/10470970.
- 55. Matza LS, Morlock R, Sexton C, Malley K, Feltner D. Identifying HAM-A cutoffs for mild, moderate, and severe generalized anxiety disorder. *Int J Methods Psychiatr Res.* 2010. doi:10.1002/mpr.323
- 56. Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. *J Health Soc Behav.* 1983. doi:10.2307/2136404
- 57. Stasiewicz PR, Brandon TH, Bradizza CM. Effects of extinction context and retrieval cues on renewal of alcohol-cue reactivity among alcohol-dependent outpatients. *Psychol Addict Behav*. 2007;21(2):244-248. doi:10.1037/0893-164X.21.2.244
- 58. Jatlow P, O'Malley SS. Clinical (nonforensic) application of ethyl glucuronide measurement: are we ready? *Alcohol Clin Exp Res.* 2010;34(6):968-975. doi:10.1111/j.1530-0277.2010.01171.x
- 59. Jatlow PI, Agro A, Wu R, et al. Ethyl glucuronide and ethyl sulfate assays in clinical trials, interpretation, and limitations: results of a dose ranging alcohol challenge study and 2 clinical trials. *Alcohol Clin Exp Res.* 2014;38(7):2056-2065. doi:10.1111/acer.12407
- 60. Leickly E, Skalisky J, McPherson S, Orr MF, McDonell MG. High Agreement Between Benchtop and Point-of-Care Dipcard Tests for Ethyl Glucuronide. *Ther Drug Monit*. 2017;39(4):461-462. doi:10.1097/FTD.000000000000012
- 61. Yoon JH, Higgins ST, Heil SH, Sugarbaker RJ, Thomas CS, Badger GJ. Delay Discounting Predicts Postpartum Relapse to Cigarette Smoking Among Pregnant Women. *Exp Clin Psychopharmacol*. 2007. doi:10.1037/1064-1297.15.2.186
- 62. Weidberg S, Landes RD, López-Núñez C, et al. Contingency management effects on delay discounting among patients receiving smoking cessation treatment. *Psicothema*. 2015;27(4). doi:10.7334/psicothema2015.184
- 63. Yoon JH, Higgins ST, Bradstreet MP, Badger GJ, Thomas CS. Changes in the relative reinforcing effects of cigarette smoking as a function of initial abstinence. *Psychopharmacology (Berl)*. 2009. doi:10.1007/s00213-009-1541-4
- 64. Weidberg S, Landes RD, López-Núñez C, et al. Contingency management effects on delay discounting among patients receiving smoking cessation treatment. *Psicothema*. 2015. doi:10.7334/psicothema2015.184
- 65. Yoon JH, De La Garza R, Newton TF, et al. A Comparison of Mazur's k and Area Under the Curve for Describing Steep Discounters. *Psychol Rec.* 2017. doi:10.1007/s40732-017-0220-9
- 66. Ross EL, Yoon JH, Mahoney JJ, Omar Y, Newton TF, De La Garza R. The impact of self-reported life stress on current impulsivity in cocaine dependent adults. *Prog Neuro-Psychopharmacology Biol Psychiatry*. 2013. doi:10.1016/j.pnpbp.2013.06.002

IRB NUMBER: HSC-MS-18-0922 UTHealth IRB APPROVAL DATE: 05/08/2019

- 67. Weidberg S, Landes RD, García-Rodríguez O, Yoon JH, Secades-Villa R. Interaction effect of contingency management and sex on delay-discounting changes among treatment-seeking smokers. *Exp Clin Psychopharmacol*. 2015. doi:10.1037/pha0000043
- 68. García-Rodríguez O, Secades-Villa R, Weidberg S, Yoon JH. A systematic assessment of delay discounting in relation to cocaine and nicotine dependence. *Behav Processes*. 2013. doi:10.1016/i.beproc.2013.07.007
- 69. Weidberg S, Garciá-Rodríguez O, Yoon JH, Secades-Villa R. Interaction of Depressive Symptoms and Smoking Abstinence on Delay Discounting Rates. *Psychol Addict Behav.* 2015. doi:10.1037/adb0000073
- 70. Yoon JH, Higgins ST. Turning k on its head: Comments on use of an ED50 in delay discounting research. *Drug Alcohol Depend.* 2008. doi:10.1016/j.drugalcdep.2007.12.011
- 71. Secades-Villa R, Weidberg S, García-Rodríguez O, Fernández-Hermida JR, Yoon JH. Decreased delay discounting in former cigarette smokers at one year after treatment. *Addict Behav*. 2014. doi:10.1016/j.addbeh.2014.03.015
- 72. Garcia-Bueno B, Perez-Nievas BG, Leza JC. Is there a role for the nuclear receptor PPARgamma in neuropsychiatric diseases? *Int J Neuropsychopharmacol*. 2010. doi:10.1017/S1461145710000970
- 73. Miller BW, Willett KC, Desilets AR. Rosiglitazone and Pioglitazone for the Treatment of Alzheimer's Disease. *Ann Pharmacother*. 2011. doi:10.1345/aph.1Q238
- 74. Kaiser CC, Shukla DK, Stebbins GT, et al. A pilot test of pioglitazone as an add-on in patients with relapsing remitting multiple sclerosis. *J Neuroimmunol*. 2009. doi:10.1016/j.jneuroim.2009.04.011
- 75. Lovallo W. The cold pressor test and autonomic function: a review and integration. *Psychophysiology*. 1975;12(3):268-282. http://www.ncbi.nlm.nih.gov/pubmed/1153632.
- 76. McRae AL, Saladin ME, Brady KT, Upadhyaya H, Back SE, Timmerman MA. Stress reactivity: biological and subjective responses to the cold pressor and Trier Social stressors. *Hum Psychopharmacol*. 2006;21(6):377-385. doi:10.1002/hup.778
- 77. Schwabe L, Haddad L, Schachinger H. HPA axis activation by a socially evaluated cold-pressor test. *Psychoneuroendocrinology*. 2008;33(6):890-895. doi:10.1016/j.psyneuen.2008.03.001
- 78. Velasco M, Gomez J, Blanco M, Rodriguez I. The cold pressor test: pharmacological and therapeutic aspects. *Am J Ther*. 1997;4(1):34-38. http://www.ncbi.nlm.nih.gov/pubmed/10423589.
- 79. Dias NR, Schmitz JM, Rathnayaka N, et al. Anti-saccade error rates as a measure of attentional bias in cocaine dependent subjects. *Behav Brain Res.* 2015;292:493-499. doi:10.1016/j.bbr.2015.07.006
- 80. Vujanovic AA, Wardle MC, Liu S, Dias NR, Lane SD. Attentional Bias in Adults with Cannabis Use Disorders: Preliminary Data on a New Experimental Paradigm . *J Addict Dis*.

